CLINICAL TRIAL: NCT06653374
Title: "Condiciones Perinatales Que Influyen en la Morbimortalidad y atención Medica en Neonatos Del Hospital Gineco Obstétrico Isidro Ayora, Enero 2008-diciembre 2022"
Brief Title: Perinatal Conditions Influencing Morbidity, Mortality, and Medical Care in Newborns
Acronym: UCE
Status: Completed | Type: Observational
Sponsor: HOSPITAL GINECO OBSTETRICO ISIDRO AYORA (Other)
Collaborators: Universidad Central del Ecuador (Other)
Responsible Party: Principal Investigator, Santiago Vasco-Morales, Principal Investigator, HOSPITAL GINECO OBSTETRICO ISIDRO AYORA
Other Study IDs: 009-DOC-FCM-2023; 009-DOC-FCM-2023 (Other: Universidad Central del Ecuador)
Record Dates: First submitted 2024-10-01; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Preterm Birth; Low Birth Weight; Intrauterine Growth Restriction (IUGR); Perinatal Asphyxia; Neonatal Sepsis; Respiratory Distress Syndrome (RDS); Neonatal Jaundice; Congenital Malformations; Neonatal Hypoglycemia; Gestational Diabetes Mellitus (GDM); Placental Abruption; Preterm Premature Rupture of Membranes (PPROM); Hypertension, Pregnancy-Induced; Pre-Eclampsia
Keywords: Infant, Premature; Infant, Low Birth Weight; Fetal Growth Retardation; Asphyxia Neonatorum; Sepsis, Neonatal; Respiratory Distress Syndrome, Newborn; Jaundice, Neonatal; Congenital Abnormalities; Hypoglycemia, Neonatal; Hypertension, Pregnancy-Induced; Diabetes, Gestational; Placental Abruption; Premature Rupture of Fetal Membranes
MeSH Terms: conditions — Premature Birth; Fetal Growth Retardation; Neonatal Sepsis; Respiratory Distress Syndrome; Jaundice, Neonatal; Congenital Abnormalities; Diabetes, Gestational; Abruptio Placentae; Preterm Premature Rupture of the Membranes; Hypertension, Pregnancy-Induced; Pre-Eclampsia; Asphyxia Neonatorum; Respiratory Distress Syndrome, Newborn; Hypoglycemia; Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infant, Premature: The "Infant, Premature" group includes neonates born before 37 weeks of gestation at the Isidro Ayora Obstetric-Gynecologic Hospital. This cohort is particularly vulnerable to a range of complications, including respiratory distress syndrome, intraventricular hemorrhage, and infections, which are major contributors to neonatal morbidity and mortality.
  Interventions: Behavioral: Infant, Premature
- Neonatal Morbidity and Mortality Cohort: This cohort includes all live-born neonates delivered at the Isidro Ayora Obstetric-Gynecologic Hospital between January 2008 and December 2022. The study focuses on evaluating the influence of various perinatal and neonatal conditions on morbidity and mortality outcomes. Interventions of interest include obstetric management strategies (e.g., use of antenatal corticosteroids, mode of delivery), neonatal resuscitation protocols, NICU admission criteria, and the implementation of specific neonatal care practices such as early surfactant administration, infection control measures, and nutritional support.
  Interventions: Behavioral: Infant, Premature

INTERVENTIONS:
Behavioral: Infant, Premature — This intervention is distinct as it focuses specifically on observational monitoring and evaluation of neonatal outcomes without applying a therapeutic or procedural treatment. Unlike other interventional studies, the emphasis is on analyzing standard care practices, risk factor exposures (e.g., prematurity, maternal complications), and their impact on neonatal morbidity and mortality. The intervention involves systematic data collection and longitudinal follow-up to identify patterns and associations, rather than introducing new clinical techniques or treatment

SUMMARY:
This study focuses on understanding the conditions that affect newborn health and survival from pregnancy to the first weeks of life at the Isidro Ayora Hospital. The investigators will review data from 2008 to 2022 to identify key factors that may contribute to complications, help improve medical care, and reduce risks for newborns. By doing so, we aim to provide better support to families, healthcare providers, and ensure safer births.

DETAILED DESCRIPTION:
This research investigates the impact of various perinatal conditions-such as maternal health, prenatal complications, delivery methods, and neonatal management-on morbidity and mortality rates in newborns treated at the Isidro Ayora Obstetric-Gynecologic Hospital. Using a retrospective cohort design, the study analyzes data from 2008 to 2022 to identify patterns and correlations between perinatal factors and neonatal outcomes, aiming to inform evidence-based clinical practices and enhance neonatal care protocols.

Key aspects include evaluating the influence of gestational age, birth weight, maternal comorbidities (e.g., hypertension, diabetes), and obstetric complications on the health of neonates. Outcomes of interest include NICU admissions, length of hospital stay, and incidence of conditions such as respiratory distress syndrome, sepsis, and neonatal mortality. Findings will contribute to improving resource allocation, optimizing care strategies, and potentially guiding policy decisions to reduce adverse neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born at the Isidro Ayora Obstetric-Gynecologic Hospital between January 2008 and December 2022.
* Live-born neonates with complete medical records in the hospital's perinatal database.
* Neonates whose mothers received antenatal care and delivered at the hospital. Availability of maternal and neonatal data, including gestational age, birth weight, and outcome information.

Exclusion Criteria:

* Neonates with incomplete or missing medical records.
* Neonates born outside the hospital and referred postnatally.
* Stillbirths and pregnancies terminated due to maternal or fetal indications.
* Neonates discharged to other facilities immediately after birth without follow-up data in the hospital's database.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population includes all live-born neonates delivered at the Isidro Ayora Obstetric-Gynecologic Hospital between January 2008 and December 2022. The cohort encompasses neonates born to mothers of diverse socioeconomic backgrounds, varying maternal health conditions, and different obstetric risk profiles. The study focuses on evaluating neonatal outcomes based on gestational age, birth weight, and the presence of perinatal complications, such as maternal hypertension, diabetes, or preterm labor. This population represents a high-risk group typical of a tertiary care referral center, allowing for a comprehensive analysis of factors influencing neonatal morbidity and mortality.
Sampling Method: Probability Sample
Enrollment: 26000 (Actual)
Dates: Start 2023-11-12 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Neonatal Mortality Rate | first 28 days of life
  The proportion of neonates who die within the first 28 days of life out of the total number of live births.

SECONDARY OUTCOMES:
Neonatal Morbidity Incidence | first 28 days of life
  Incidence of major neonatal morbidities, including sepsis, respiratory distress syndrome, intraventricular hemorrhage, necrotizing enterocolitis, and perinatal asphyxia.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Gineco Obstétrico Isidro Ayora, Quito, Pichincha, Ecuador

IPD SHARING:
Plan to Share IPD: Undecided
The database contains sensitive information on neonates and their mothers, protected by ethical and confidentiality regulations. Due to the nature of the data and hospital policies, IPD will not be shared publicly to safeguard patient privacy and comply with local regulations. Aggregated results will be available in scientific publications, but individual data will not be accessible to third parties.